CLINICAL TRIAL: NCT03678207
Title: The Effectiveness of a Preoperative Blood Pressure Screening Program to Identify Undiagnosed Hypertension in Ambulatory Surgery Patients
Acronym: Peri-op HTN
Status: Withdrawn | Type: Observational
Why Stopped: The investigator no longer desires to persue the trial. No enrollments were made.
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0914
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2019-10

CONDITIONS: Hypertension; Perioperative Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Potential Undiagnosed HTN
  Interventions: Other: Anesthesiologist phone call

INTERVENTIONS:
Other: Anesthesiologist phone call — Patients receiving ambulatory surgery with no prior diagnosis of hypertension but have elevated blood pressure prior to surgery. Patients will receive a phone call from a participating anesthesiologist 1-3 days after surgery notifying them of their high blood pressure and obtaining oral consent to participate in the study. Patients will receive reminders via mail about following up with their PCP.

SUMMARY:
Elevated blood pressure is the largest contributing risk factor to all-cause and cardiovascular mortality. According to the U.S. Preventive Services Task Force, hypertension affects nearly 30% of the adult population. Many patients remain undiagnosed, despite the consensus that screening and timely diagnosis is paramount. In this study, 108 ambulatory surgery patients with elevated blood pressure (160/90) that are not yet formally diagnosed with hypertension will be enrolled and alerted of their high blood pressure by a co-investigator MD. They will request permission to follow-up with the patient and the patient's primary care provider 6 months after the initial phone call to check in on the status of their diagnosis and any action taken (lifestyle changes, medication) to alleviate their high blood pressure. Patients will receive a follow-up letter/email at 6 and 3 months to remind them of their potential diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective ambulatory surgery
* Patients with a pre-operative elevated BP defined as greater than 160/90
* Patients above the age of 18
* English speaking

Exclusion Criteria:

* Patients with a pre-existing diagnosis of HTN
* Patients who are taking a hypertensive medication
* Patients who had a pre-operative surgical screening assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving elective ambulatory surgery with a preoperative blood pressure measurement greater than 160 (systolic) and/or 90 (diastolic)
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Diagnosis of hypertension 6 months after surgery | 6 months postoperative
  The number of patients with previously undiagnosed hypertension that have obtained a formal diagnosis of hypertension

SECONDARY OUTCOMES:
PCP follow up 6 months after surgery | 6 months postoperative
  Number of patients that followed-up with a primary care physician for further hypertension testing within 6 months of surgery
Hypertension treatment 6 months after surgery | 6 months postoperative
  Number of patients that followed-up for their hypertension that received some sort of treatment, either medication or lifestyle

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No